CLINICAL TRIAL: NCT02778815
Title: The Development and Initial Evaluation of a Web-based, Compassion-focussed Course for New Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canterbury Christ Church University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IsobelGammerMRP2015
Record Dates: First submitted 2016-05-16; First posted 2016-05-20 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: New Mothers' Well-being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kindness for Mums (Experimental): An online self-help course designed to promote self-kindness and self-compassion in new mothers
  Interventions: Other: Kindness for Mums
- Wait list control (No Intervention): A waiting list control group, who will receive access to the online self-help intervention once the RCT is complete.

INTERVENTIONS:
Other: Kindness for Mums
  Arms: Kindness for Mums

SUMMARY:
This study examines the relationship between self-compassion and wellbeing in new mothers and whether an online self-help course for new mothers can help to improve their wellbeing and self-compassion.

DETAILED DESCRIPTION:
This study is a randomised controlled trial (RCT) comparing an online self-help course ('Kindness for Mums') with a wait-list control. A battery of self-report measures will be administered online at baseline (week 0), post-intervention (week 6) and at follow-up (week 12). Baseline data will also be used to examine the relationship between self-compassion and wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* New mothers (can be biological, adoptive or full-time foster mother)
* Able to complete baseline measures when infant aged 0-12 months
* Fluent in English
* Live in the United Kingdom
* Able to access the internet

Exclusion Criteria:

* Experiencing suicidal ideation at the time of enrolment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2016-09; Primary Completion 2017-05-11 (Actual); Study Completion 2017-05-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline at 6-weeks on the Warwick-Edinburgh Mental Well-Being Scale | Post-intervention (i.e. 6-weeks after baseline)

SECONDARY OUTCOMES:
Change from baseline at 6-weeks on the Self-Compassion Scale | Post-intervention (i.e. 6 weeks post baseline)
Change from baseline at 6-weeks on the Forms of Self-Criticising/Attacking and Self-Reassuring Scale | Post-intervention (i.e. 6 weeks post baseline)
Change from baseline at 6-weeks on the Depression, Anxiety and Stress Scale 21-item version | Post-intervention (i.e. 6 weeks post baseline)
Change from baseline at 12-weeks on the Warwick-Edinburgh Mental Well-Being Scale | 12-weeks after baseline
Change from baseline at 12-weeks on the Self-Compassion Scale | 12-weeks after baseline
Change from baseline at 12-weeks on the Forms of Self-Criticising/Attacking and Self-Reassuring Scale | 12-weeks after baseline
Change from baseline at 12-weeks on the Depression, Anxiety and Stress Scale 21-item version | 12-weeks after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Isobel Gammer, BA, MSc, Principal Investigator — Canterbury Christ Church University

IPD SHARING:
Plan to Share IPD: No